CLINICAL TRIAL: NCT05862519
Title: A Single-Group, Open-Label Clinical Study to Evaluate the Efficacy of Four Supplements on Improving Readiness for Intimacy
Brief Title: A Clinical Study to Evaluate the Efficacy of Four Supplements on Improving Readiness for Intimacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: 906 CMVI Holdings (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20287
Record Dates: First submitted 2023-04-20; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Libido; Intimacy; Gastrointestinal Issues

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants will begin taking the Reset supplement for 5 days. Then there will be a 2-day break with no products taken (wash out period).
  Participants will then begin taking the following 2 supplements: Stay Ready Fiber and libido with a partial overlap of products.
  Stay Ready Fiber will be taken from day 7 through 21, three capsules will be taken twice daily in the morning and afternoon.
  Libido will be taken from day 7 through 28, 2 capsules will be taken daily, preferably with a meal.
  Participants will then begin taking the Testosterone supplement. Testosterone will be taken from day 28 through to 84, 2 capsules will be taken daily, preferably with a meal.
  Interventions: Dietary Supplement: Reset; Dietary Supplement: Stay Ready Fiber; Dietary Supplement: Libido; Dietary Supplement: Testosterone supplement

INTERVENTIONS:
Dietary Supplement: Reset — Pure for Men Reset is a Vegan, Proprietary Blend of Toxin Eliminating Cleanser: Cascara Sagrada Bark, Senna Leaf, Psyllium Husk, Licorice Root, and Aloe Vera Gel. Taken on Day 1 to Day 5.
  Other Names: Pure for Men Reset Supplement
Dietary Supplement: Stay Ready Fiber — Stay Ready Fiber is a Vegan, 100% Natural, Proprietary Blend of Digestive Aids: Psyllium Husk, Aloe Vera Extract, Chia Seeds & Flaxseed. Taken from Day 7 through Day 21.
  Other Names: Pure for Men Stay Ready Fiber Capsules
Dietary Supplement: Libido — Supplement designed to support endurance and increased arousal. Contains L-Citrulline, L-Arginine and Black Pepper Fruit Extract (Piper Nigrum). Taken from Day 7 through to Day 28.
  Other Names: Pure for Men Pump Enhancer
Dietary Supplement: Testosterone supplement — Supplement designed to enhance testosterone production. Contains Ashwagandha, Zinc, Vitamin D, Maca, and Tongkat Ali. Taken from Day 28 through Day 84.
  Other Names: Pure for Men T-Support

SUMMARY:
This study is to evaluate the efficacy of four supplements designed to help participants get ready for sexual intimacy through improving digestion, weight management, sexual drive and stamina, and physical endurance during workouts and overall mood and quality of life. This study will be conducted as a single group, virtual trial, in which all participants will take all four supplements and complete online questionnaires. Participants will take the indicated supplements for the indicated amounts of time over 12 weeks. Questionnaires will be completed at baseline, and then at indicated times throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male (biological at birth) within the LGBTQIA+ community
* Aged between 18-44
* Generally healthy - don't live with any uncontrolled chronic disease
* Generally active lifestyle or seeking to achieve health improvement
* Sexually active with a partner

Exclusion Criteria:

* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Anyone with known severe allergic reactions.
* Unwilling to follow the study protocol.
* Currently experiencing significant symptoms of a mental disorder that might interfere with study participation (e.g. eating disorder, obsessive-compulsive disorder, posttraumatic stress syndrome, bipolar disorder)
* Current substance abuse disorder
* Diagnosis of an autoimmune disease, such as multiple sclerosis and rheumatoid arthritis
* Self-reported or diagnosed high blood pressure or hypotension (BP < 90 over 60)
* Currently, or in the past 6 months, undergoing hormone therapy
* Any medical condition that is unstable or uncontrolled
* A history of sexual trauma or abuse
* Has introduced any new prescription medication or supplements within the past 12 weeks that influence gastrointestinal issues, libido, or testosterone production.

Ages: 18 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-06-06 (Estimated); Study Completion 2023-06-13 (Estimated)

PRIMARY OUTCOMES:
Changes in subject's perception of readiness and confidence for intimacy, and sex drive/arousal [Time Frame: Baseline to 12 weeks] | 12 weeks
  Survey-based assessment (0-5 scale) of changes in reduction in preparation time for intimacy, sexual arousal, and sexual endurance.

SECONDARY OUTCOMES:
Changes in digestion, stamina and endurance during workouts, overall confidence, mood and quality of life [Time Frame: Baseline to 12 weeks] | 12 weeks
  Survey-based assessment (0-5 scale) of changes in digestion, stamina and endurance during workouts, overall confidence, mood and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States